CLINICAL TRIAL: NCT01523145
Title: CopenHeartRFA - A Randomized Clinical Trial Investigating the Effect and Meaning of Integrated Rehabilitation Versus Usual Follow-up of Patients Treated for Atrial Fibrillation With Radio Frequency Ablation
Brief Title: CopenHeartRFA - Integrated Rehabilitation of Patients Treated for Atrial Fibrillation With Radio Frequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHCopenHeartRFA
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Radio Frequency Ablation; Rehabilitation; Physical capacity; Quality of life; Integrated rehabilitation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rehabilitation; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Rehabilitation
- Control gruop (Experimental)
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Rehabilitation — Integrated Rehabilitation consisting of exercise training (minimum 3 times a week for a total of twelve weeks) and psychoeducational care (4 sessions over 6 months)
  Arms: Intervention
Other: Control Group — usual follow-up Standard follow-up at the participating heart center
  Arms: Control gruop

SUMMARY:
Atrial fibrillation is the most common arrhythmia and affect 1-2 % of the population in the western world. Atrial fibrillation can be treated with a relatively new procedure, called radiofrequency ablation.

The aim of this study is to explore if patients treated with ablation for atrial fibrillation, benefit from an integrated rehabilitation programme, that consist of physical training and psycho-educative consultations with a specialised nurse.

The hypothesis is, that integrated rehabilitation can improve mental health, physical capacity and other factors.

DETAILED DESCRIPTION:
1-2 % of the population in the western world live with atrial fibrillation. One way to treat atrial fibrillation is with radiofrequency ablation. Ablation is a relatively new treatment and therefore only few studies has been exploring how the patients are doing after discharge. In Denmark the patients are not offered rehabilitation, only brief follow-up with a doctor. Therefore the aim of this study is to explore if the patients will benefit from a integrated rehabilitation programme consisting of physical training and psycho-educational intervention.

A randomized clinical trial is conducted to investigate the effect and meaning of an integrated rehabilitation programme on the physical and psychosocial functioning of patients treated for atrial fibrillation with radiofrequency ablation. The trial is a parallel arm design.

A mixed methods embedded experimental design is chosen to include both quantitative and qualitative data to evaluate the intervention. The intervention consists of four psycho-educational consultations provided by specialized nurses and a twelve week individualized exercise training programme provided by physiotherapists. A qualitative post-intervention study will explore rehabilitation participation experiences.

The hypothesis is, that integrated rehabilitation can improve mental health, physical capacity, self-rated health, quality of life, sleep-quality and reduce anxiety, depression, health care utilisation, work cessation and mortality in patients treated for atrial fibrillation with radiofrequency ablation and that it is cost effective.

210 patients will be included.

Questionnaires, cardiopulmonary testing, 6 minute walking test and qualitative interviews will be used to evaluate the effect and meaning of the programme.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* treated for atrial fibrillation with radiofrequency ablation on Rigshospitalet, Denmark
* 18 years or older
* speaking and understanding Danish
* providing written informed consent

Exclusion Criteria:

* unable to understand study instructions
* who are pregnant or breastfeeding
* with considerable illness in the musculoskeletal system or with physical disability, which complicates exercise training
* who does strenuous physical training several times a week on competition level
* who does not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in physical capacity | 1, 4 and 12 months
  Measured by Peak VO2 via ergospirometry testing

SECONDARY OUTCOMES:
Change in mental component scale | 1, 4, 6, 12 and 24 months
  Measured by the mental component scale (MCS) in the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Signe S Risom, RN, MSc, Principal Investigator — Rigshospitalet, Denmark; Selina K Berg, MScN, ph.d., Principal Investigator — Copenhagen University Hospital Rigshospitalet, University Hospital Gentofte; Ann-Dorthe O Zwisler, MD, ph.d., Principal Investigator — Copenhagen University Hospital Rigshospitalet, National Institute of Public Health, University of Southern Denmark; Jesper H Svendsen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Risom SS, Zwisler AD, Sibilitz KL, Rasmussen TB, Taylor RS, Thygesen LC, Madsen TS, Svendsen JH, Berg SK. Cardiac Rehabilitation for Patients Treated for Atrial Fibrillation With Ablation Has Long-Term Effects: 12-and 24-Month Follow-up Results From the Randomized CopenHeartRFA Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1877-1886. doi: 10.1016/j.apmr.2020.06.026. Epub 2020 Aug 1. PMID 32750373
- [Derived] Risom SS, Lind J, Dickson VV, Berg SK. Exploring the Mechanism of Effectiveness of a Psychoeducational Intervention in a Rehabilitation Program (CopenHeartRFA) for Patients Treated With Ablation for Atrial Fibrillation: A Mixed Methods Study. J Cardiovasc Nurs. 2019 Jul/Aug;34(4):336-343. doi: 10.1097/JCN.0000000000000584. PMID 31058705
- [Derived] Risom SS, Zwisler AD, Rasmussen TB, Sibilitz KL, Svendsen JH, Gluud C, Hansen JL, Winkel P, Thygesen LC, Perhonen M, Hansen J, Dunbar SB, Berg SK. The effect of integrated cardiac rehabilitation versus treatment as usual for atrial fibrillation patients treated with ablation: the randomised CopenHeartRFA trial protocol. BMJ Open. 2013 Feb 20;3(2):e002377. doi: 10.1136/bmjopen-2012-002377. Print 2013. PMID 23430599